CLINICAL TRIAL: NCT04279964
Title: Engaging Practices and Communities in the Development of Interventions to Promote HPV Vaccine Uptake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-0338; 1R21CA230878-01A1 (NIH)
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Primary Prevention
Keywords: Immunization; Boot Camp Translation; Adolescent; Human Papillomavirus; Vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Boot Camp Translation (Experimental): Intervention practices will undergo the Boot Camp Translation process.
  Interventions: Behavioral: Boot Camp Translation
- Control (Active Comparator): Control practice will behave as usual.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Boot Camp Translation — Practices in the intervention arm will participate in the Boot Camp Translation process, where BCT Community Advisory group members will come together to develop and implement practice relevant materials to promote adolescent vaccination.
  Arms: Boot Camp Translation
Other: Control — No intervention. Practices will continue to behave as usual.
  Arms: Control

SUMMARY:
The overarching goal of this project is to implement Boot Camp Translation (BCT) methodology to translate the guidelines and evidence for human papillomavirus (HPV) vaccine into a practice and provider level intervention designed to improve its acceptability and uptake.

DETAILED DESCRIPTION:
As a community engagement approach, Boot Camp Translation (BCT), is a 6-9-month iterative process that brings together multiple stakeholders, including patients, parents, and community members, to translate evidence-based guidelines and recommendations into locally relevant and meaningful messages, materials, and programs.

Aim 1: Implement BCT in three geographically distinct Colorado communities to translate the current evidence for HPV vaccination into locally relevant interventions designed to increase vaccine uptake.

Aim 2: Evaluate the impact of the BCT- designed intervention on practice-level HPV vaccination initiation rates.

The long-term goal is to develop a replicable approach and low-cost method of increasing HPV vaccine uptake that is easily adaptable to different settings and sociodemographic contexts.

ELIGIBILITY:
Inclusion Criteria:

All child patients who have received health supervision at participating practices during the 12 month prior to intervention and the 12 month following intervention implementation, who are ages 9-26 years, and whose parents have not requested removal from the Colorado Immunization Information System (CIIS) will be eligible for the assessment of practice immunization rates in the pre and post periods.

Exclusion Criteria:

* No subjects will be excluded because of gender, ethnicity, or insurance status.
* Any child whose parents have requested removal from the immunization registry; any child with hypersensitivity to any component of one of the recommended vaccines; any child who has moved to a primary care provider other than one at the study clinics.

Ages: 9 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2400 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Initiation of HPV vaccination series, 9-17 | Up to 12 months
  Percent of 9-17 year olds who have received >=1 dose of the HPV vaccine by September 29, 2021

SECONDARY OUTCOMES:
Differences in initiation rates between intervention vs. control, 9-10 | 12 months
  Comparison of boys vs. girls who have received >1=dose of HPV vaccine by September 29, 2021
Differences in initiation rates between intervention vs. control, 11-12 | 12 months
  Comparison of boys vs. girls who have received >1=dose of HPV vaccine by September 29, 2021
Differences in initiation rates between intervention vs. control, 13-17 | 12 months
  Comparison of boys vs. girls who have received >1=dose of HPV vaccine by September 29, 2021
Differences in initiation rates between intervention vs. control, 18-26 | 12 months
  Percent of 18-26 year olds who have received >=1 dose of the HPV vaccine by September 29, 2021

CONTACTS AND LOCATIONS:
Overall Officials: Sean O'Leary, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brewer SE, Simpson MJ, Rice JD, Skenadore A, O'Leary ST. Engaging practices and communities in the development of interventions to promote HPV vaccine uptake: a protocol for implementing Boot Camp Translation in the private practice setting. BMJ Open. 2020 Dec 12;10(12):e041685. doi: 10.1136/bmjopen-2020-041685. PMID 33310806

DOCUMENTS (1):
  • Informed Consent Form (2021-07-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT04279964/ICF_000.pdf